CLINICAL TRIAL: NCT00936091
Title: Effects of Vitamin A Supplementation on Intestinal Parasitic Reinfections, Growth, Iron Status and Educational Achievement Among Orang Asli Schoolchildren in Pos Betau, Pahang, Malaysia
Brief Title: Effects of Vitamin A Supplementation on Intestinal Parasitic Reinfections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Collaborators: University of Malaya (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Prof. Dr. Johari Surin, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PS178-2007B, PS178-2007B
Record Dates: First submitted 2009-07-03; First posted 2009-07-09 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-07

CONDITIONS: Intestinal Parasitic Infections; Malnutrition; Anemia
Keywords: intestinal parasitic infections; malnutrition; Anemia
MeSH Terms: conditions — Malnutrition; Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): 125 schoolchildren were allocated randomly to receive placebo
  Interventions: Drug: Placebo
- vitamin A supplement (Active Comparator): 125 children received vitamin A supplements capsules (200 000 IU)
  Interventions: Drug: vitamin A supplements

INTERVENTIONS:
Drug: vitamin A supplements — gelatinous and reddish opaque capsules containing 200 000 IU vitamin A
  Other Names: Group B
  Arms: vitamin A supplement
Drug: Placebo — 125 children received placebo capsules
  Other Names: Group A
  Arms: placebo

SUMMARY:
Intestinal parasitic infections, malnutrition and iron deficiency anaemia (IDA) are still considered as public health problems in rural Malaysia especially among Orang Asli children. Despite intermittent control programmes, the prevalence of these problems is still high suggesting the need of other control and interventions measures. This randomized double-blind, placebo-controlled trial was carried out among Orang Asli schoolchildren from Sekolah Kebangsaan Betau in Pos Betau, Pahang (200 km northeast Kuala Lumpur) to investigate the effects of vitamin A supplementation on intestinal parasitic reinfections, growth, iron status and educational achievement.

HYPOTHESES

1. Vitamin A supplementation has a negative effect on intestinal parasitic reinfections and the worm burden of infections among Orang Asli schoolchildren in Pos Betau, Kuala Lipis, Pahang.
2. Vitamin A supplementation has a positive effect on growth (weight and height) among Orang Asli schoolchildren.
3. Vitamin A supplementation is effective in improving serum iron status among Orang Asli schoolchildren.
4. Vitamin A supplementation has a positive effect on cognitive function and educational achievement among Orang Asli schoolchildren.

DETAILED DESCRIPTION:
Children from Sekolah Kebangsaan Betau in Pos Betau, Kuala Lipis, Pahang served as the target population for this study.

The selection criteria for study subjects were the following:

* Age 7-12 years (according to birth date in birth certificate).
* Non-menstruating females (age <13)
* No history or evidence of underlying haematological-related diseases such as thalassaemia and ovalocytosis.
* No evidence of concomitant severe and/or chronic illness such as acute respiratory tract infections, mental retardation and neurological deficits.
* Consent of parent to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-12 years (according to birth date in birth certificate).
* No evidence of concomitant severe and/or chronic illness such as acute respiratory tract infections, mental retardation and neurological deficits.
* Consent of parent to participate in the study.

Exclusion Criteria:

* history or evidence of underlying haematological-related diseases such as thalassaemia and ovalocytosis.
* menstruating females (age >13)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
intestinal parasitic infections | 6 months

SECONDARY OUTCOMES:
growth , iron status & educational achievement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M Al-Mekhlafi, PhD, Principal Investigator — University of Malaya
Locations (1):
- National school of Pos Betau, Kuala Lipis, Pahang, Malaysia

REFERENCES:
- [Background] Donnen P, Brasseur D, Dramaix M, Vertongen F, Zihindula M, Muhamiriza M, Hennart P. Vitamin A supplementation but not deworming improves growth of malnourished preschool children in eastern Zaire. J Nutr. 1998 Aug;128(8):1320-7. doi: 10.1093/jn/128.8.1320. PMID 9687551
- [Background] Hadi H, Stoltzfus RJ, Dibley MJ, Moulton LH, West KP Jr, Kjolhede CL, Sadjimin T. Vitamin A supplementation selectively improves the linear growth of indonesian preschool children: results from a randomized controlled trial. Am J Clin Nutr. 2000 Feb;71(2):507-13. doi: 10.1093/ajcn/71.2.507. PMID 10648265
- [Background] Payne LG, Koski KG, Ortega-Barria E, Scott ME. Benefit of vitamin A supplementation on ascaris reinfection is less evident in stunted children. J Nutr. 2007 Jun;137(6):1455-9. doi: 10.1093/jn/137.6.1455. PMID 17513406
- [Background] Tanumihardjo SA, Permaesih D, Muhilal. Vitamin A status and hemoglobin concentrations are improved in Indonesian children with vitamin A and deworming interventions. Eur J Clin Nutr. 2004 Sep;58(9):1223-30. doi: 10.1038/sj.ejcn.1601953. PMID 15054437
- [Derived] Al-Mekhlafi HM, Anuar TS, Al-Zabedi EM, Al-Maktari MT, Mahdy MA, Ahmed A, Sallam AA, Abdullah WA, Moktar N, Surin J. Does vitamin A supplementation protect schoolchildren from acquiring soil-transmitted helminthiasis? A randomized controlled trial. Parasit Vectors. 2014 Aug 15;7:367. doi: 10.1186/1756-3305-7-367. PMID 25127885